CLINICAL TRIAL: NCT05758818
Title: A Randomized, Positive and Placebo-Controlled Trial to Evaluate the Effects of Milademetan Administration on Cardiac Repolarization in Healthy Subjects
Brief Title: A Study of Milademetan Administration on Cardiac Repolarization in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RAIN-3258
Record Dates: First submitted 2023-01-29; First posted 2023-03-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Repolarization
MeSH Terms: interventions — Moxifloxacin; milademetan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A = Placebo (negative control) (Placebo Comparator): Dosage Form: Capsules
  Route of Administration: Oral
  The placebo and milademetan will be identical in appearance.
  Interventions: Drug: Placebo
- B = Moxifloxacin (positive control) (Active Comparator): Dosage Form: Tablets
  Route of Administration: Oral
  Dosage: 400 mg
  Interventions: Drug: Moxifloxacin (positive control)
- C = Milademetan (Experimental): Drug: Milademetan
  Dosage:
  Part 1: 300, 330, 360 mg. Part 2: 260 mg single oral dose or higher, as determined in Part 1.
  Interventions: Drug: Milademetan

INTERVENTIONS:
Drug: Placebo — Participants will receive a single dose of placebo on Day 1, Day 8 or Day 15 of part 2
  Arms: A = Placebo (negative control)
Drug: Moxifloxacin (positive control) — Participants will receive a single dose of moxifloxacin on Day 1,Day 8, or Day 15 of Part 2
  Arms: B = Moxifloxacin (positive control)
Drug: Milademetan — Participants will receive a single dose of Milademetan on Day 1 for part 1
  Participants will receive a single dose of milademetan on Day 1, Day 8, or Day 15 of Part 2
  Arms: C = Milademetan

SUMMARY:
This will be a Phase 1, single-center, 2-part study in healthy subjects. Parts 1 and 2 need to be conducted in sequential order.

DETAILED DESCRIPTION:
Part 1 will enroll up to 3 cohorts of 6 healthy adult subjects to receive a single dose. The total duration of participation from the Screening visit to the follow-up will be up to 7 weeks (up to 45 days).

Part 2 of this study will randomize approximately 32 subjects. The total duration of participation from the Screening visit to the follow-up will be up to 8 weeks (up to 55 days).

ELIGIBILITY:
Inclusion Criteria:

1. Is capable of understanding informed consent and is willing and able to provide written informed consent.
2. Is willing to comply with all protocol procedures.
3. Healthy, male, nonsmoking (for at least 90 days) subjects from 18 through 55 years of age, inclusive, at Screening, and healthy, female, nonsmoking (for at least 90 days) subjects of nonchildbearing potential from 18 through 55 years of age, inclusive, at Screening.
4. Body weight > 50 kg, body mass index between 18.0 and 30 kg/m2, inclusive.

Exclusion Criteria:

1. Past or present clinically relevant systemic disease as judged by the Investigator including, but not limited to, clinically relevant medical abnormalities such as psychiatric, neurologic, pulmonary, respiratory, cardiac, gastrointestinal, genitourinary, renal, hepatic, metabolic, endocrinologic, hematological, or autoimmune disorders making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study in the opinion of the Investigator.
2. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
3. Knowledge of any kind of cardiovascular disorder/condition/procedure known to increase the possibility of QT prolongation or a history of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, hypomagnesemia, congenital long QT syndrome, or family history of long QT syndrome, or Brugada syndrome), or cardiac conduction disorders.
4. Resting supine systolic blood pressure greater than 140 mm Hg; resting supine diastolic blood pressure greater than 90 mm Hg at Screening or Day -1. Blood pressure measurements may be repeated once at the discretion of the Investigator.
5. Resting supine HR less than 45 beats per minute or greater than 100 beats per minute at Screening or Day -1 (may be repeated once at the discretion of the Investigator). Minor deviations are acceptable if considered to be of no clinical significance by the Investigator.
6. Abnormal 12-lead ECG at Screening or Day -1 (a single repeat is allowed), including:

   1. QTcF > 450 msec
   2. QRS > 110 msec
   3. PR > 200 msec
   4. Second or third-degree atrioventricular block
7. Any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant at Screening or Day -1.
8. Dosing in another clinical trial within the last 30 days (or 5 half-lives, whichever is longer) prior to Day -1.
9. Family history of unexplainable sudden death at < 50 years of age.
10. History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations, clinically significant head injury, or near drowning with hospital admission.
11. Known allergic reactions to moxifloxacin (for Part 2 only) or any study medication or history of tendonitis or tendon rupture as a result of moxifloxacin or any other quinolone type drug use (for Part 2 only).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Part 1:Up to 15 days
  The intensity of all AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Number of participants with adverse events (AEs) | Part 2: Up to 25 days
  The intensity of all AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Incidence of laboratory abnormalities based on hematology test results | Part 1:Up to 15 days
  Hematocrit, Hemoglobin, Mean cell hemoglobin
Incidence of laboratory abnormalities based on hematology test results | Part 2: Up to 25 days
  Hematocrit, Hemoglobin, Mean cell hemoglobin
Incidence of laboratory abnormalities based on clinical chemistry test results | Part 1:Up to 15 days
  Alanine aminotransferase, Albumin, Alkaline phosphatase, Aspartate aminotransferase
Incidence of laboratory abnormalities based on clinical chemistry test results | Part 2: Up to 25 days
  Alanine aminotransferase, Albumin, Alkaline phosphatase, Aspartate aminotransferase
Incidence of laboratory abnormalities based on urinalysis test results | Part 1:Up to 15 days
  Bilirubin, color and appearance, glucose, ketones, protein
Incidence of laboratory abnormalities based on urinalysis test results | Part 2: Up to 25 days
  Bilirubin, color and appearance, glucose, ketones, protein
Vital signs measurements | Part 1:Up to 15 days
  Supine systolic blood pressure in mmHg and supine diastolic blood pressure in mmHg
Vital signs measurements | Part 2: Up to 25 days
  Supine systolic blood pressure in mmHg and supine diastolic blood pressure in mmHg
Change from baseline in QT interval of the ECG | Part 1:Up to 15 days
  QT interval measured in msec
Change from baseline in QT interval of the ECG | Part 2: Up to 25 days
  QT interval measured in msec

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | Part 1:Up to 15 days
  observed maximum plasma concentration in ng/ml
Observed maximum plasma concentration (Cmax) | Part 2: Up to 25 days
  observed maximum plasma concentration in ng/ml
Time to observed maximum concentration (Tmax) | Part 1:Up to 15 days
  time to observed maximum concentration in hour
Time to observed maximum concentration (Tmax) | Part 2: Up to 25 days
  time to observed maximum concentration in hour
area under the time-concentration curve from time zero to the time of the last quantifiable concentration (AUC0-tlast) | Part 1:Up to 15 days
  Expressed as ng/ml x hr
area under the time-concentration curve from time zero to the time of the last quantifiable concentration (AUC0-tlast) | Part 2: Up to 25 days
  Expressed as ng/ml x hr

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No